CLINICAL TRIAL: NCT00476775
Title: Ethnic Dance and Screen Time Reduction to Prevent Weight Gain in Latina Girls
Acronym: ECHALE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DK073006 (NIH); SPO 33483 (Other: Stanford University); R01DK073006 (NIH)
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Obesity; Overweight; Excessive Weight Gain
Keywords: obesity; prevention; girls; Latina/Hispanic; Dance; television; screen time
MeSH Terms: conditions — Obesity; Overweight | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- After school ethnic dance and home-based screen time reduction (Experimental): After school ethnic dance classes and home-based screen time reduction intervention
  Interventions: Behavioral: after school ethnic dance program - ballet folklorica; Behavioral: culturally-tailored, home-based screen time reduction
- Health and Nutrition Education (Active Comparator): Health and nutrition education active placebo control intervention
  Interventions: Behavioral: culturally-tailored health and nutrition education

INTERVENTIONS:
Behavioral: after school ethnic dance program - ballet folklorica
  Arms: After school ethnic dance and home-based screen time reduction
Behavioral: culturally-tailored, home-based screen time reduction
  Arms: After school ethnic dance and home-based screen time reduction
Behavioral: culturally-tailored health and nutrition education
  Arms: Health and Nutrition Education

SUMMARY:
A randomized controlled trial to test the efficacy of an after school ethnic dance program plus a culturally-tailored, home-based screen time reduction intervention to reduce weight gain (body mass index) among lower socioeconomic status, pre-adolescent Latina girls.

DETAILED DESCRIPTION:
We propose a 2-arm, parallel group, randomized controlled trial to test the efficacy of an after school ethnic dance program plus a culturally-tailored, home-based screen time reduction intervention to reduce weight gain (body mass index) among lower socioeconomic status, pre-adolescent Latina girls. The control group will receive an "active-placebo" information-based health education intervention. A total of 240 7-9 year old girls will be randomized to the two conditions, and both interventions will last for the full 2-year period of the study for each girl.

Latina girls are at increased risk of obesity and obesity-related morbidities. However, effective and generalizable obesity prevention programs for this rapidly growing population are not available. After school ethnic dance programs are highly motivating, and an innovative approach to providing a large "dose" of moderate-to-vigorous physical activity for Latina girls. After school programs may also indirectly reduce sedentary behavior and improve diet. Dance is fun for pre-adolescent girls, it plays an important social and cultural role in Latino communities, and after school dance classes are a potentially generalizable "environmental" intervention strategy. Our past pilot studies and ongoing trials of ethnic dance interventions demonstrate that (1) dance is a highly attractive and feasible form of activity for pre-adolescent girls and (2) a dance intervention can result in reduced weight gain (BMI) and increased fitness among girls.

Latina girls are also heavy consumers of screen-based media, television, videotapes/DVDs and video games. Excessive screen time is considered one of the most modifiable causes of childhood obesity. We propose a culturally-tailored, home-based screen time reduction intervention, delivered by bilingual, Latina, Community Health Advisors (CHAs). Our prior and ongoing studies demonstrate the feasibility and potential efficacy of (1) reducing children's screen time to reduce weight gain and (2) providing home-based behavior change interventions to low-income Latino families using CHAs. All interventions will be further developed, revised, and pilot-tested with Latina girls and their families through formative research.

240 girls Latina girls will be recruited over 18 months from six public elementary schools serving low-income Latino communities in northern CA. Measures will be collected in girls' homes at baseline, 6, 12, 18 and 24 months, including height and weight, waist circumference, triceps skinfold thickness, blood pressure and resting heart rate, physical activity monitoring by accelerometry, media use, 24-hour dietary recalls, weight concerns, depressive symptoms, school performance, sexual maturation, and demographics. Body Mass Index (BMI) is the primary outcome measure. The primary outcome analysis will compare individual trajectories of change in BMI in the treatment and control groups over the entire two-year course of the trial, using random regression models. The study is powered (90%) to detect a clinically-significant effect. Specific Aims include:

1. To test the efficacy of a combined, after school ethnic dance and home-based screen time reduction intervention to reduce weight gain (BMI) over 2 years.

   Primary hypothesis: Compared to controls, girls in the treatment group will significantly reduce their weight gain (BMI) over the two-year study period.
2. To test the effects of a combined, after school ethnic dance and home-based screen time reduction intervention on secondary outcomes over two years.

   Secondary hypotheses: Compared to controls, girls in the treatment group will significantly reduce their waist circumference, triceps skinfold thickness, systolic and diastolic resting blood pressures, resting heart rate, television, videotape/DVD and video game use, meals eaten with TV, daily dietary energy intake, percent of energy from fat, weight concerns and depressive symptoms, and significantly increase their daily physical activity, daily moderate to vigorous physical activity, liking for physical activity, and school performance.
3. To evaluate potential demographic, cultural, psychological, and biological moderators and mediators of intervention effects on BMI and secondary outcomes, to evaluate correlates and risk factors for change in BMI and secondary outcomes, and to evaluate intervention delivery variables and their relationships to outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Defined as Latina or Hispanic by parent/guardian.
* Attends one of the participating public elementary schools.

Exclusion Criteria:

* Diagnosed with a medical condition affecting growth.
* Taking medications affecting growth.
* A condition limiting participation in the interventions.
* A condition limiting participation in the assessments.
* Plan to move from the area within the next 24 months.

Ages: 7 Years to 9 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 233 (Actual)
Dates: Start 2007-05; Primary Completion 2011-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | change over 2 years

SECONDARY OUTCOMES:
waist circumference | over 2 years
triceps skinfold thickness | over 2 years
systolic and diastolic resting blood pressures | over 2 years
resting heart rate | over 2 years
screen time | over 2 years
meals eaten with television | over 2 years
average dietary energy intake and percent of energy from fat | over 2 years
average daily total physical activity and moderate-to-vigorous physical activity | over 2 years
weight concerns | over 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N Robinson, M.D., M.P.H., Principal Investigator — Stanford University
Locations (1):
- Stanford Prevention Research Center, Stanford, California, United States